CLINICAL TRIAL: NCT03946618
Title: Human Safety and Feasibility Study of Neurophysiologically Based Brain State Tracking and Modulation in Focal Epilepsy
Brief Title: Neurophysiologically Based Brain State Tracking and Modulation in Focal Epilepsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Medtronic (Industry)
Responsible Party: Principal Investigator, Gregory Worrell, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 18-005483; UH2NS095495-03 (NIH)
Record Dates: First submitted 2019-04-19; First posted 2019-05-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Epilepsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Epilepsy (Experimental): Patients with dominant temporal lobe epilepsy and bilateral temporal lobe epilepsy
  Interventions: Device: Medtronic Summit System, Olympus

INTERVENTIONS:
Device: Medtronic Summit System, Olympus — Electrical brain stimulation with an implantable pulse generator

SUMMARY:
Researchers are trying to determine if tracking seizure occurrence, seizure probability, behavioral state, cognition, and mood can be achieved using an implantable brain sensing and stimulation device (Medtronic RC+S Summit) coupled to an external, handheld, patient assistant device (PAD) with capability for patient interaction (patient data input). The system (RC+S & PAD) provides intracranial EEG (iEEG) sensing, electrical brain stimulation, and machine learning algorithms running on the RC+S and PAD that will be coupled with electrical brain stimulation (EBS) to prevent seizures and improve quality of life in patients with epilepsy.

DETAILED DESCRIPTION:
This study will include patients with dominant temporal lobe epilepsy and bilateral temporal lobe epilepsy. The plan is to have 10 patients take part in this study at Mayo Clinic Rochester.

ELIGIBILITY:
Inclusion Criteria

* Focal epilepsy, including seizures with and without impairment of consciousness, and secondarily generalized seizures:

  * Disabling seizure counts >3 per month (Disabling seizures are those with significant negative impact on the patients life)
  * Drug resistance to >2 appropriate seizure drugs with therapeutic serum concentrations
  * Not a good candidate for resective surgery or at significant risk for verbal memory decline as determined by our institution's multidisciplinary Epilepsy Surgery Committee.
  * For 3 months prior to enrollment, subject's anti-seizure medication dosages have been stable and subject has had at least 6 disabling (as defined in Inclusion Criteria 1) seizures per month, on average, with a seizure-free interval not to exceed 30 days. Seizures must be separated by a minimum of eight hours not to be considered part of a cluster. A cluster of seizures, for the purpose of this criterion, shall be considered a single seizure.
* With the exception of epilepsy, subject must be medically and neurologically stable.
* Mayo Clinic Epilepsy Surgery Committee approval for brain stimulation therapy obtained on clinical grounds and without reference to this protocol.
* Age 18 to 75
* Ability and willingness to provide informed consent and participate in the study protocol. Subject is able to interpret and to respond, in accordance with the study protocol, to the advisory indicators provided by the device.
* Subject has seizures that are distinct, stereotypical events that can be reliably counted by the patient or caregiver.
* Subject can reasonably be expected to maintain a seizure diary alone or with the assistance of a competent individual.
* Subject is able to complete regular office visits and telephone appointments in accordance with the study protocol requirements.
* A female subject must have a negative serum pregnancy test within two weeks prior to entering the study, and, if sexually active, must be using a reliable form of birth control, be surgically sterile, or be at least two years post-menopausal.
* Subject's seizure focus, based upon clinical semiology, intracranial electroencephalographic (iEEG) findings, and/or neuroimaging, shall demonstrate bilateral medial temporal lobe epilepsy or unilateral temporal lobe epilepsy of dominant temporal lobe origin.
* Subject has been informed of his or her eligibility for resective surgery as a potential alternative to the study, if such surgery is a reasonable option.
* Subject speaks and reads English.
* Subject has had a brain magnetic resonance imaging (MRI) epilepsy evaluation within the past two years.
* Subject has iEEG documentation of ictal events consistent with his or her predominant current seizure type.
* Subject's anatomy will permit implantation of the Medtronic Investigational RC+S generator within 20 mm of the skin surface.
* Subject can reasonably be expected to periodically check battery levels and recharge devices (Implanted neural stimulator (INS), Clinical Telemetry Module (CTM), and EPAD tablet) alone or with the assistance of a competent individual.

Exclusion Criteria

* For 3 months prior to enrollment, subject's anti-seizure medication dosages have not been stable, or subject has had more than 25 disabling (as defined in Inclusion Criteria 1) seizures per month, on average, or there was a seizure-free interval longer than 30 days within the past 3 months. Clinical seizures must be separated by a minimum of eight hours to not be considered part of a cluster. Cluster seizures are considered a single seizure event.
* Subject has a contraindication to magnetic resonance imaging.
* Subject has a substance abuse history (alcohol, prescription, or illicit medications) within the preceding two years.
* Subject participated in another drug or device trial within the preceding 30 days.
* Subject has been hospitalized for a psychiatric condition within the preceding two years or has had a history of psychosis within the preceding two years (excluding post-ictal psychosis).
* Subject is implanted with pacemaker, implantable cardiac defibrillator, cardiac management product, or a medical device that interferes with the RC+S device. This includes, but is not limited to, direct brain neurostimulators, spinal cord stimulators, vagus nerve stimulators (VNS), and cochlear implants. Patients with a vagus nerve stimulator implanted but turned off through the duration of the study may be enrolled, provided their clinical status has been stable for at least one month with VNS turned off. Alternatively, patients with a VNS may have the previously disabled VNS removed at time of surgery to implant the Medtronic RC+S.
* Subject has been diagnosed with psychogenic or non-epileptic seizures.
* Subject has been diagnosed with primary generalized seizures.
* Subject has experienced unprovoked status epilepticus in the preceding year.
* Subject has had therapeutic surgery to treat epilepsy that may interfere with electrode placement.
* Subject is on anticoagulants and is unable to discontinue them peri-surgically, as required by the neurosurgeon or Investigator.
* Subject has significant platelet dysfunction from medical conditions or medications (including, particularly, aspirin or sodium valproate). If platelet dysfunction is suspected, subject can be enrolled only if a hematologist, the Investigator, and the neurosurgeon judge it to be advisable.
* Subject is ineligible for cranial surgery.
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE) experienced with the RC+S system | Through 15 months
  Number of AEs reported
24/7 continuous iEEG monitoring | Through 15 months
  Number of RC+S systems that generates continues 24/7 EEG without interruption
Change in mood | Baseline, biweekly for up to 15 months
  Measured using daily mood and anxiety trackers questionnaire, where 1 is not at all and 7 is extremely
Change in anxiety | Baseline, biweekly for up to 15 months
  Measured using anxiety Generalized Anxiety Disorder 7-item (GAD-7) scale, where 0 is not at all sure and 3 is nearly every day
Tracking cognition | Baseline, biweekly for up to 15 months
  Measured using free recall task

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Worrell, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balzekas I, Trzasko J, Yu G, Richner TJ, Mivalt F, Sladky V, Gregg NM, Van Gompel J, Miller K, Croarkin PE, Kremen V, Worrell GA. Method for cycle detection in sparse, irregularly sampled, long-term neuro-behavioral timeseries: Basis pursuit denoising with polynomial detrending of long-term, inter-ictal epileptiform activity. PLoS Comput Biol. 2024 Apr 25;20(4):e1011152. doi: 10.1371/journal.pcbi.1011152. eCollection 2024 Apr. PMID 38662736